CLINICAL TRIAL: NCT01418014
Title: Adolescent Master Protocol
Acronym: AMP
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Tulane University School of Medicine (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); NIH Office of AIDS Research (OAR) (NIH)
Responsible Party: Principal Investigator, Paige Williams, Senior Lecturer on Biostatistics, Harvard School of Public Health (HSPH)
Other Study IDs: HD052102 - PH200; PH200 (Other: PHACS Protocol Number)
Record Dates: First submitted 2011-07-22; First posted 2011-08-16 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, cell pellets, plasma, saliva, and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infected Cohort: Perinatally HIV-infected adolescents from 7 years of age (7th birthday) up to but not including the 16th birthday at enrollment, engaged in care with ART treatment history available.
- Uninfected Cohort: HIV-uninfected adolescents from 7 years of age (7th birthday) up to but not including the 16th birthday at enrollment born to HIV-infected mothers.

SUMMARY:
The advances in treatment to prevent maternal HIV transmission to neonates have been groundbreaking. As a result, the number of new perinatally-infected children in the U.S. is now small. Subsequent improvements in the treatment of HIV-infected infants and children have been equally remarkable, ensuring that most previously infected American children have survived and are approaching adolescence. In addition, the number of HIV-infected adolescents worldwide is growing substantially in both resource-poor countries and in countries with increasing levels of health care. Therefore, there is a global cohort of children who have been living with HIV infection since birth who are aging into adolescence. Little is definitively known about the impact of HIV infection and its treatment on the maturation process in these children.

AMP is a prospective cohort study designed to define the impact of HIV infection and antiretroviral therapy on pre-adolescents and adolescents with perinatal HIV infection. Domains to be investigated include growth and sexual maturation, metabolic risk factors for cardiovascular disease, cardiac function, bone health, neurologic, neurodevelopment, language, hearing and behavioral function, and sexually transmitted infections (STI).

DETAILED DESCRIPTION:
The primary objectives of AMP are:

1. To define the impact of HIV infection and ART on growth and pubertal development (and their hormonal regulation), along with the cognitive, academic, and social development, of pre-adolescents and adolescents with perinatal HIV infection as they move through adolescence into adulthood.
2. To identify infectious and non-infectious complications of HIV disease, including the toxicities of antiretroviral therapy (ART).
3. To investigate:

   * Cognitive and behavioral changes over time, including medication adherence, family and social function, and high risk behaviors such as risky sexual behavior, licit and illicit drug use, and alcohol use;
   * Changes in language and hearing;
   * Changes in glucose metabolism, body composition, and bone mineralization;
   * Changes in lipid metabolism and other risk factors for cardiovascular disease;
   * Risk factors for secondary transmission of HIV; and
   * The occurrence and clinical course of cervical HPV infections among females.

The domain-specific aims of AMP are:

1. Growth and sexual maturation: To longitudinally track growth and sexual maturation and the factors that influence growth and maturation in HIV-infected children when compared to HIV-exposed but uninfected children.
2. Metabolic risk factors for cardiovascular disease: To characterize the emergence of abnormal glucose metabolism, lipid abnormalities, body composition and other risk factors for cardiovascular disease and identify the contributing influences in HIV-infected children when compared to HIV-exposed but uninfected children.
3. Cardiac function: To estimate the prevalence of cardiac structural and functional abnormalities in HIV-infected children and youth when compared to HIV-exposed but uninfected children.
4. Bone mineral density: To estimate the differences in bone mineral density of HIV-infected children when compared to HIV-exposed but uninfected children and to identify factors contributing to abnormal bone mineralization.
5. Neurologic, neurodevelopment, language, and behavioral function:

   * To examine cognitive and behavioral outcomes of HIV-infected children and adolescents, including high risk behaviors such as risky sexual behavior, licit and illicit drug use, and alcohol use, neurodevelopmental impairment, school achievement and to compare them with an HIV-exposed but uninfected control cohort.
   * To examine non-adherence to antiretroviral therapy and predictors of non-adherence among HIV-infected children receiving ART.
   * To examine family and psychosocial factors associated with emotional and behavioral problems.
6. Adolescent gynecology and STI infection:

   * To evaluate the incidence of and risk factors for acquiring STIs/vaginal infections (C. trachomatis, N. gonorrhea, T. vaginalis, syphilis, genital warts, HPV, and HSV) for males and females, and in addition bacterial vaginosis for females.
   * To evaluate the incidence, predictors, and outcomes of pregnancy.

ELIGIBILITY:
HIV-Infected Cohort

Inclusion Criteria:

* Perinatal HIV infection as documented in the medical record.
* Age 7 years (7th birthday) up to but not including the 16th birthday at enrollment.
* Engaged in care and ART history is available.
* Either: Previous or current enrollment in any of the studies included on the list of approved studies allowing for enrollment into AMP as specified in the protocol. Children participating in other studies may be enrolled with approval of the Protocol Team. Additional approved protocols are listed on the PHACS website; Or: Available medical record documentation since birth of 1)ART exposure history 2)Opportunistic Infection (OI) prophylaxis exposure history 3) Viral load and CD4 count history and 4) Major medical events history
* Willingness to participate and provide parental/legal guardian permission with assent. Children who do not know their HIV infection status will not be excluded.

Exclusion criteria: HIV acquired by other than maternal-child transmission (e.g., blood products, sexual contact, and IV drug use) as documented in the medical record.

HIV-Uninfected, HIV-Exposed Control Cohort

Inclusion criteria:

* HIV-uninfected and born to an HIV-infected mother as documented in the medical record.
* Age 7 years (7th birthday) up to but not including the 16th birthday at enrollment.
* Previous or current enrollment in any of the studies included on the list of approved studies allowing for enrollment into AMP. Children participating in other studies may be enrolled with approval of the Protocol Team. Additional approved protocols will be listed on the PHACS website; Or: Available medical record documentation since birth of 1)ART exposure history and 2) Major medical events history.
* Willingness to participate and provide parental/legal guardian permission with assent.

Exclusion Criteria: None.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected and -uninfected children from 7 years of age (7th birthday) up to but not including the 16th birthday at the time of enrollment born to HIV-infected mothers. Participants will be children previously enrolled in any of the studies included on the list of approved studies for co-enrollment (see below) or has medical record documentation since birth of key medical data related to their HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 678 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Abnormal growth | Annually for 10 years
  Assessed via measurement of height, weight, skinfold thickness, mid-upper arm and waist and hip circumference, nutrition and physical activity questionnaires ; subjects meeting growth trigger based on height measurements also have the following laboratory assessments: IGF-I, IGFBP-3, and GHBP. A growth hormone stimulation test may also be required at the recommendation of the endocrinologist.
Delayed sexual maturation | Annually for 10 years except if subject reaches Tanner Stage 5
  Assessed via tanner staging; subjects meeting the growth trigger based on the results of the tanner staging will also have the following laboratory assessments: morning LH, FSH, estradiol, and testosterone
Abnormal bone mineral density | Two DXAs, two years apart, per HIV-infected subject; one DXA per uninfected subject; X-ray at same time as DXA unless subject Tanner Stage 5
  Assessed via DXA scan and x-ray for bone age; subjects meeting the BMD trigger based on the DXA also have the following laboratory assessments: TSH, calcium, 25-hydroxy-vitamin D, bone-specific alkaline, N-terminal telopeptide of type I collagen phosphatase, and PTH in real time and repository specimens for assay of pro-inflammatory cytokines (IL-1, IL-6, TNF-a)
Dyslipidemia | Annually for 10 years
  Assessed via lipid testing; subjects meeting the metabolic trigger based on the results of the lipid tests also have the following measurements: endothelial dysfunction (I, E, P-selectins: V, I-CAM-1, endothelin-1, hs-CRP, homocysteine, apolipoprotein B, lipoprotein (a), and vWF antigen)
Cardiac abnormalities | Measured once per subject until study reached 400 echocardiograms
  Assessed through the administration of echocardiograms and serum biomarkers (ProBNP)
Hearing dysfunction | Once per subject.
  Assessed via audiologic evaluation conducted by an audiologist.
Language dysfunction | Annually for 10 years
  Assessed using the Woodcock and CELF IV language tests
Neurodevelopmental abnormalities | Annually for 10 years
  Assessed via the following neurodevelopmental tests: WISC IV, WAIS IV, BRIEF, Children's Color Trails Test, Trail Making Tests, WIAT-II screen, ABAS, Parent Child Relationship Inventory, BASC-2, Quality of Life Interview, Stressful Life Events Questionnaire, Monitoring the Future
Substance Use | Annually starting at a minimum of 10 years of age for 10 years
  The assessment of sexual activity is conducted using an Audio Computer Assisted Survey Instrument (ACASI). ACASI uses computer and voice recordings so that the participant hears (through headphones) and sees (on the screen) each question and response list. The use of ACASI is proven to minimize response bias due to the presence of an interviewer.
Sexual Activity | Annually starting at a minimum of 10 years of age for 10 years
  The assessment of substance use is conducted using an Audio Computer Assisted Survey Instrument (ACASI). ACASI uses computer and voice recordings so that the participant hears (through headphones) and sees (on the screen) each question and response list. The use of ACASI is proven to minimize response bias due to the presence of an interviewer.
Pregnancy | Annually for 10 years
  Assessed via medical record review to record incidents of pregnancy
Sexually Transmitted Infection | Annually for 10 years
  Assessed via medical record review to record results of clinically conducted STI and Pap testing and pelvic exams
Mitochondrial dysfunction | Annually for 10 years
  Assessed via measurement of serum lactate levels, OXPHO immunoassays, mitochondrial specific oxidative stress, mtDNA copies/cell, mrRNA transcripts
Lactic acidosis | Annually for 10 years
  Assessed through the measurement of blood lactate levels using a point-of-care lactate measuring device; a single venous lactate measurement will be conducted in cases where the POC lactate measure is elevated
Renal abnormalities | Annually for 10 years
  Assessed through the following laboratory measurements: chemistry panel, urinalysis, protein/creatinine ratio, dip stick urine test

CONTACTS AND LOCATIONS:
Overall Officials: Paige L Williams, Principal Investigator — Harvard School of Public Health (HSPH); Russell Van Dyke, M.D., Principal Investigator — Tulane University School of Medicine
Locations (15):
- United States (14):
  - University of California San Diego, La Jolla, California
  - University of Colorado Denver Health Sciences Center, Aurora, Colorado
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Rutgers - New Jersey Medical School, Newark, New Jersey
  - Bronx Lebanon Hospital Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
- San Juan Research Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Kapetanovic S, Leister E, Nichols S, Miller T, Tassiopoulos K, Hazra R, Gelbard HA, Malee KM, Kammerer B, Mendez AJ, Williams PL; Pediatric HIV/AIDS Cohort Study Team. Relationships between markers of vascular dysfunction and neurodevelopmental outcomes in perinatally HIV-infected youth. AIDS. 2010 Jun 19;24(10):1481-91. doi: 10.1097/QAD.0b013e32833a241b. PMID 20539091
- [Result] Van Dyke RB, Patel K, Siberry GK, Burchett SK, Spector SA, Chernoff MC, Read JS, Mofenson LM, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study. Antiretroviral treatment of US children with perinatally acquired HIV infection: temporal changes in therapy between 1991 and 2009 and predictors of immunologic and virologic outcomes. J Acquir Immune Defic Syndr. 2011 Jun 1;57(2):165-73. doi: 10.1097/QAI.0b013e318215c7b1. PMID 21407086
- [Result] Siberry GK, Patel K, Van Dyke RB, Hazra R, Burchett SK, Spector SA, Paul ME, Read JS, Wiznia A, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study(PHACS). CD4+ lymphocyte-based immunologic outcomes of perinatally HIV-infected children during antiretroviral therapy interruption. J Acquir Immune Defic Syndr. 2011 Jul 1;57(3):223-9. doi: 10.1097/QAI.0b013e318218e068. PMID 21423022
- [Result] Malee KM, Tassiopoulos K, Huo Y, Siberry G, Williams PL, Hazra R, Smith RA, Allison SM, Garvie PA, Kammerer B, Kapetanovic S, Nichols S, Van Dyke R, Seage GR 3rd, Mellins CA; Pediatric HIV/AIDS Cohort Study Team. Mental health functioning among children and adolescents with perinatal HIV infection and perinatal HIV exposure. AIDS Care. 2011 Dec;23(12):1533-44. doi: 10.1080/09540121.2011.575120. PMID 21702707
- [Result] Mellins CA, Tassiopoulos K, Malee K, Moscicki AB, Patton D, Smith R, Usitalo A, Allison SM, Van Dyke R, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study. Behavioral health risks in perinatally HIV-exposed youth: co-occurrence of sexual and drug use behavior, mental health problems, and nonadherence to antiretroviral treatment. AIDS Patient Care STDS. 2011 Jul;25(7):413-22. doi: 10.1089/apc.2011.0025. Epub 2011 May 5. PMID 21992620
- [Result] Geffner ME, Patel K, Miller TL, Hazra R, Silio M, Van Dyke RB, Borkowsky W, Worrell C, DiMeglio LA, Jacobson DL; Pediatric HIV/AIDS Cohort Study. Factors associated with insulin resistance among children and adolescents perinatally infected with HIV-1 in the pediatric HIV/AIDS cohort study. Horm Res Paediatr. 2011;76(6):386-91. doi: 10.1159/000332957. Epub 2011 Oct 26. PMID 22042056
- [Result] Jacobson DL, Patel K, Siberry GK, Van Dyke RB, DiMeglio LA, Geffner ME, Chen JS, McFarland EJ, Borkowsky W, Silio M, Fielding RA, Siminski S, Miller TL; Pediatric HIV/AIDS Cohort Study. Body fat distribution in perinatally HIV-infected and HIV-exposed but uninfected children in the era of highly active antiretroviral therapy: outcomes from the Pediatric HIV/AIDS Cohort Study. Am J Clin Nutr. 2011 Dec;94(6):1485-95. doi: 10.3945/ajcn.111.020271. Epub 2011 Nov 2. PMID 22049166
- [Result] Miller TI, Borkowsky W, DiMeglio LA, Dooley L, Geffner ME, Hazra R, McFarland EJ, Mendez AJ, Patel K, Siberry GK, Van Dyke RB, Worrell CJ, Jacobson DL; Pediatric HIV/AIDS Cohort Study (PHACS); Shearer W, Cooper N, Harris L, Purswani M, Baig M, Cintron A, Puga A, Navarro S, Patton D, Burchett S, Karthas N, Kammerer B, Yogev R, Malee K, Hunter S, Cagwin E, Wiznia A, Burey M, Nozyce M, Chen J, Gobs E, Grant M, Knapp K, Allison K, Garvie P, Acevedo-Flores M, Rios H, Olivera V, Silio M, Borne C, Sirois P, Spector S, Norris K, Nichols S, McFarland E, Barr E, Chambers C, Watson D, Messenger N, Belanger R, Dieudonne A, Bettica L, Adubato S, Scott G, Himic L, Willen E. Metabolic abnormalities and viral replication are associated with biomarkers of vascular dysfunction in HIV-infected children. HIV Med. 2012 May;13(5):264-75. doi: 10.1111/j.1468-1293.2011.00970.x. Epub 2011 Dec 4. PMID 22136114
- [Result] Torre P 3rd, Zeldow B, Hoffman HJ, Buchanan A, Siberry GK, Rice M, Sirois PA, Williams PL; Pediatric HIVAIDS Cohort Study. Hearing loss in perinatally HIV-infected and HIV-exposed but uninfected children and adolescents. Pediatr Infect Dis J. 2012 Aug;31(8):835-41. doi: 10.1097/INF.0b013e31825b9524. PMID 22549437
- [Result] Rice ML, Buchanan AL, Siberry GK, Malee KM, Zeldow B, Frederick T, Purswani MU, Hoffman HJ, Sirois PA, Smith R, Torre P 3rd, Allison SM, Williams PL. Language impairment in children perinatally infected with HIV compared to children who were HIV-exposed and uninfected. J Dev Behav Pediatr. 2012 Feb;33(2):112-23. doi: 10.1097/DBP.0b013e318241ed23. PMID 22179050
- [Result] Siberry GK, Leister E, Jacobson DL, Foster SB, Seage GR 3rd, Lipshultz SE, Paul ME, Purswani M, Colin AA, Scott G, Shearer WT. Increased risk of asthma and atopic dermatitis in perinatally HIV-infected children and adolescents. Clin Immunol. 2012 Feb;142(2):201-8. doi: 10.1016/j.clim.2011.10.005. Epub 2011 Oct 30. PMID 22094294
- [Result] Smith R, Chernoff M, Williams PL, Malee KM, Sirois PA, Kammerer B, Wilkins M, Nichols S, Mellins C, Usitalo A, Garvie P, Rutstein R; Pediatric HIV/AIDS Cohort Study (PHACS) Team. Impact of HIV severity on cognitive and adaptive functioning during childhood and adolescence. Pediatr Infect Dis J. 2012 Jun;31(6):592-8. doi: 10.1097/INF.0b013e318253844b. PMID 22592486
- [Result] Tassiopoulos K, Moscicki AB, Mellins C, Kacanek D, Malee K, Allison S, Hazra R, Siberry GK, Smith R, Paul M, Van Dyke RB, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study. Sexual risk behavior among youth with perinatal HIV infection in the United States: predictors and implications for intervention development. Clin Infect Dis. 2013 Jan;56(2):283-90. doi: 10.1093/cid/cis816. Epub 2012 Nov 7. PMID 23139252
- [Result] DiMeglio LA, Wang J, Siberry GK, Miller TL, Geffner ME, Hazra R, Borkowsky W, Chen JS, Dooley L, Patel K, van Dyke RB, Fielding RA, Gurmu Y, Jacobson DL; Pediatric HIVAIDS Cohort Study (PHACS). Bone mineral density in children and adolescents with perinatal HIV infection. AIDS. 2013 Jan 14;27(2):211-20. doi: 10.1097/QAD.0b013e32835a9b80. PMID 23032412
- [Result] Purswani M, Patel K, Kopp JB, Seage GR 3rd, Chernoff MC, Hazra R, Siberry GK, Mofenson LM, Scott GB, Van Dyke RB; Pediatric HIVAIDS Cohort Study. Tenofovir treatment duration predicts proteinuria in a multiethnic United States Cohort of children and adolescents with perinatal HIV-1 infection. Pediatr Infect Dis J. 2013 May;32(5):495-500. doi: 10.1097/INF.0b013e31827f4eff. PMID 23249917
- [Result] Lipshultz SE, Williams PL, Wilkinson JD, Leister EC, Van Dyke RB, Shearer WT, Rich KC, Hazra R, Kaltman JR, Jacobson DL, Dooley LB, Scott GB, Rabideau N, Colan SD; Pediatric HIV/AIDS Cohort Study (PHACS). Cardiac status of children infected with human immunodeficiency virus who are receiving long-term combination antiretroviral therapy: results from the Adolescent Master Protocol of the Multicenter Pediatric HIV/AIDS Cohort Study. JAMA Pediatr. 2013 Jun;167(6):520-7. doi: 10.1001/jamapediatrics.2013.1206. PMID 23608879
- [Result] Williams PL, Abzug MJ, Jacobson DL, Wang J, Van Dyke RB, Hazra R, Patel K, Dimeglio LA, McFarland EJ, Silio M, Borkowsky W, Seage GR 3rd, Oleske JM, Geffner ME; International Maternal Pediatric and Adolescent AIDS Clinical Trials P219219C Study and the Pediatric HIVAIDS Cohort Study. Pubertal onset in children with perinatal HIV infection in the era of combination antiretroviral treatment. AIDS. 2013 Jul 31;27(12):1959-70. doi: 10.1097/QAD.0b013e328361195b. PMID 24145244
- [Result] Sharma TS, Jacobson DL, Anderson L, Gerschenson M, Van Dyke RB, McFarland EJ, Miller TL; Pediatric HIV/AIDS Cohort Study (PHACS). Short communication: The relationship between mitochondrial dysfunction and insulin resistance in HIV-infected children receiving antiretroviral therapy. AIDS Res Hum Retroviruses. 2013 Sep;29(9):1211-7. doi: 10.1089/AID.2012.0354. PMID 23742635
- [Result] Usitalo A, Leister E, Tassiopoulos K, Allison S, Malee K, Paul ME, Smith R, Van Dyke RB, Seage GR 3rd, Mellins CA. Relationship between viral load and self-report measures of medication adherence among youth with perinatal HIV infection. AIDS Care. 2014 Jan;26(1):107-15. doi: 10.1080/09540121.2013.802280. Epub 2013 Jun 26. PMID 23800360
- [Result] Alperen J, Brummel S, Tassiopoulos K, Mellins CA, Kacanek D, Smith R, Seage GR 3rd, Moscicki AB. Prevalence of and risk factors for substance use among perinatally human immunodeficiency virus-infected and perinatally exposed but uninfected youth. J Adolesc Health. 2014 Mar;54(3):341-9. doi: 10.1016/j.jadohealth.2013.09.003. Epub 2013 Nov 13. PMID 24239286
- [Result] Kapetanovic S, Griner R, Zeldow B, Nichols S, Leister E, Gelbard HA, Miller TL, Hazra R, Mendez AJ, Malee K, Kammerer B, Williams PL; Pediatric HIV/AIDS Cohort Study Team. Biomarkers and neurodevelopment in perinatally HIV-infected or exposed youth: a structural equation model analysis. AIDS. 2014 Jan 28;28(3):355-64. doi: 10.1097/QAD.0000000000000072. PMID 24670521
- [Result] Patel K, Wang J, Jacobson DL, Lipshultz SE, Landy DC, Geffner ME, Dimeglio LA, Seage GR 3rd, Williams PL, Van Dyke RB, Siberry GK, Shearer WT, Young L, Scott GB, Wilkinson JD, Fisher SD, Starc TJ, Miller TL; Pediatric HIV/AIDS Cohort Study (PHACS). Aggregate risk of cardiovascular disease among adolescents perinatally infected with the human immunodeficiency virus. Circulation. 2014 Mar 18;129(11):1204-12. doi: 10.1161/CIRCULATIONAHA.113.001978. Epub 2013 Dec 23. PMID 24366631
- [Result] Siberry GK, Patel K, Pinto JA, Puga A, Mirza A, Miller TL, Van Dyke RB; Pediatric HIVAIDS Cohort Study. Elevated aspartate aminotransferase-to-platelet ratio index in perinatally HIV-infected children in the United States. Pediatr Infect Dis J. 2014 Aug;33(8):855-7. doi: 10.1097/INF.0000000000000348. PMID 25222306
- [Result] Garvie PA, Zeldow B, Malee K, Nichols SL, Smith RA, Wilkins ML, Williams PL; Pediatric HIVAIDS Cohort Study (PHACS). Discordance of cognitive and academic achievement outcomes in youth with perinatal HIV exposure. Pediatr Infect Dis J. 2014 Sep;33(9):e232-8. doi: 10.1097/INF.0000000000000314. PMID 25361033
- [Result] IeDEA and ART Cohort Collaborations; Avila D, Althoff KN, Mugglin C, Wools-Kaloustian K, Koller M, Dabis F, Nash D, Gsponer T, Sungkanuparph S, McGowan C, May M, Cooper D, Chimbetete C, Wolff M, Collier A, McManus H, Davies MA, Costagliola D, Crabtree-Ramirez B, Chaiwarith R, Cescon A, Cornell M, Diero L, Phanuphak P, Sawadogo A, Ehmer J, Eholie SP, Li PC, Fox MP, Gandhi NR, Gonzalez E, Lee CK, Hoffmann CJ, Kambugu A, Keiser O, Ditangco R, Prozesky H, Lampe F, Kumarasamy N, Kitahata M, Lugina E, Lyamuya R, Vonthanak S, Fink V, d'Arminio Monforte A, Luz PM, Chen YM, Minga A, Casabona J, Mwango A, Choi JY, Newell ML, Bukusi EA, Ngonyani K, Merati TP, Otieno J, Bosco MB, Phiri S, Ng OT, Anastos K, Rockstroh J, Santos I, Oka S, Somi G, Stephan C, Teira R, Wabwire D, Wandeler G, Boulle A, Reiss P, Wood R, Chi BH, Williams C, Sterne JA, Egger M. Immunodeficiency at the start of combination antiretroviral therapy in low-, middle-, and high-income countries. J Acquir Immune Defic Syndr. 2014 Jan 1;65(1):e8-16. doi: 10.1097/QAI.0b013e3182a39979. PMID 24419071
- [Result] Persaud D, Patel K, Karalius B, Rainwater-Lovett K, Ziemniak C, Ellis A, Chen YH, Richman D, Siberry GK, Van Dyke RB, Burchett S, Seage GR 3rd, Luzuriaga K; Pediatric HIV/AIDS Cohort Study. Influence of age at virologic control on peripheral blood human immunodeficiency virus reservoir size and serostatus in perinatally infected adolescents. JAMA Pediatr. 2014 Dec;168(12):1138-46. doi: 10.1001/jamapediatrics.2014.1560. PMID 25286283
- [Result] Torre P 3rd, Yao TJ, Zeldow B, Williams P, Hoffman HJ, Siberry GK; Pediatric HIVAIDS Cohort Study (PHACS). Distortion product otoacoustic emission data in perinatally HIV-infected and HIV-exposed but uninfected children and adolescents in the Pediatric HIV/AIDS Cohort Study. Pediatr Infect Dis J. 2015 Mar;34(3):276-8. doi: 10.1097/INF.0000000000000598. PMID 25742077
- [Result] Crowell CS, Huo Y, Tassiopoulos K, Malee KM, Yogev R, Hazra R, Rutstein RM, Nichols SL, Smith RA, Williams PL, Oleske J, Muller WJ; PACTG 219C Study Team and the Pediatric HIVAIDS Cohort Study (PHACS). Early viral suppression improves neurocognitive outcomes in HIV-infected children. AIDS. 2015 Jan 28;29(3):295-304. doi: 10.1097/QAD.0000000000000528. PMID 25686678
- [Result] Krogstad P, Patel K, Karalius B, Hazra R, Abzug MJ, Oleske J, Seage GR 3rd, Williams PL, Borkowsky W, Wiznia A, Pinto J, Van Dyke RB; Pediatric HIVAIDS Cohort Study, IMPAACT 219C, and NICHD International Site Development Initiative (NISDI) Investigators. Incomplete immune reconstitution despite virologic suppression in HIV-1 infected children and adolescents. AIDS. 2015 Mar 27;29(6):683-93. doi: 10.1097/QAD.0000000000000598. PMID 25849832
- [Result] Nichols SL, Brummel SS, Smith RA, Garvie PA, Hunter SJ, Malee KM, Kammerer BL, Wilkins ML, Rutstein R, Tassiopoulos K, Chernoff MC, Mellins CA; Pediatric HIVAIDS Cohort Study. Executive Functioning in Children and Adolescents With Perinatal HIV Infection. Pediatr Infect Dis J. 2015 Sep;34(9):969-75. doi: 10.1097/INF.0000000000000809. PMID 26376309
- [Result] Uban KA, Herting MM, Williams PL, Ajmera T, Gautam P, Huo Y, Malee KM, Yogev R, Csernansky JG, Wang L, Nichols SL, Sowell ER; Pediatric HIVAIDS Cohort and the Pediatric Imaging, Neurocognition, and Genetics Studies. White matter microstructure among youth with perinatally acquired HIV is associated with disease severity. AIDS. 2015 Jun 1;29(9):1035-44. doi: 10.1097/QAD.0000000000000648. PMID 26125138
- [Result] Siberry GK, Patel K, Bellini WJ, Karalius B, Purswani MU, Burchett SK, Meyer WA 3rd, Sowers SB, Ellis A, Van Dyke RB; Pediatric HIV AIDS Cohort Study (PHACS); Pediatric HIV AIDS Cohort Study PHACS. Immunity to Measles, Mumps, and Rubella in US Children With Perinatal HIV Infection or Perinatal HIV Exposure Without Infection. Clin Infect Dis. 2015 Sep 15;61(6):988-95. doi: 10.1093/cid/civ440. Epub 2015 Jun 9. PMID 26060291
- [Result] Herting MM, Uban KA, Williams PL, Gautam P, Huo Y, Malee K, Yogev R, Csernansky J, Wang L, Nichols S, Van Dyke R, Sowell ER. Default Mode Connectivity in Youth With Perinatally Acquired HIV. Medicine (Baltimore). 2015 Sep;94(37):e1417. doi: 10.1097/MD.0000000000001417. PMID 26376381
- [Result] Fairlie L, Karalius B, Patel K, van Dyke RB, Hazra R, Hernan MA, Siberry GK, Seage GR 3rd, Agwu A, Wiznia A; Pediatric HIV AIDS Cohort Study (PHACS), The International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT). CD4+ and viral load outcomes of antiretroviral therapy switch strategies after virologic failure of combination antiretroviral therapy in perinatally HIV-infected youth in the United States. AIDS. 2015 Oct 23;29(16):2109-19. doi: 10.1097/QAD.0000000000000809. PMID 26182197
- [Result] Nichols SL, Chernoff MC, Malee K, Sirois PA, Williams PL, Figueroa V, Woods SP; Memory and Executive Functioning Substudy of the Pediatric HIVAIDS Cohort Study. Learning and Memory in Children and Adolescents With Perinatal HIV Infection and Perinatal HIV Exposure. Pediatr Infect Dis J. 2016 Jun;35(6):649-54. doi: 10.1097/INF.0000000000001131. PMID 26967812
- [Result] Agwu AL, Yao TJ, Eshleman SH, Patel K, Huang W, Burchett SK, Siberry GK, Van Dyke RB; Pediatric HIVAIDS Cohort Study. Phenotypic Coreceptor Tropism in Perinatally HIV-infected Youth Failing Antiretroviral Therapy. Pediatr Infect Dis J. 2016 Jul;35(7):777-81. doi: 10.1097/INF.0000000000001158. PMID 27078121
- [Result] Kapogiannis BG, Leister E, Siberry GK, Van Dyke RB, Rudy B, Flynn P, Williams PL; REACH Study and the PACTG 219219C Study. Prevalence of and progression to abnormal noninvasive markers of liver disease (aspartate aminotransferase-to-platelet ratio index and Fibrosis-4) among US HIV-infected youth. AIDS. 2016 Mar 27;30(6):889-98. doi: 10.1097/QAD.0000000000001003. PMID 26959353
- [Result] Fisher SD, Starc TJ, Guerra V, Williams PL, Wilkinson JD, Lipshultz SE. Declining Incidence of Systolic Left Ventricular Dysfunction in Human Immunodeficiency Virus-Infected Individuals Treated With Highly Active Antiretroviral Therapy. Am J Cardiol. 2016 Apr 1;117(7):1194-5. doi: 10.1016/j.amjcard.2016.01.008. Epub 2016 Jan 14. No abstract available. PMID 26993978
- [Result] Caniglia EC, Patel K, Huo Y, Williams PL, Kapetanovic S, Rich KC, Sirois PA, Jacobson DL, Hernandez-Diaz S, Hernan MA, Seage GR 3rd; Pediatric HIVAIDS Cohort Study. Atazanavir exposure in utero and neurodevelopment in infants: a comparative safety study. AIDS. 2016 May 15;30(8):1267-78. doi: 10.1097/QAD.0000000000001052. PMID 26867136
- [Result] Purswani MU, Patel K, Winkler CA, Spector SA, Hazra R, Seage GR 3rd, Mofenson L, Karalius B, Scott GB, Van Dyke RB, Kopp JB; Pediatric HIVAIDS Cohort Study. Brief Report: APOL1 Renal Risk Variants Are Associated With Chronic Kidney Disease in Children and Youth With Perinatal HIV Infection. J Acquir Immune Defic Syndr. 2016 Sep 1;73(1):63-8. doi: 10.1097/QAI.0000000000001010. PMID 27035887
- [Result] Van Dyke RB, Patel K, Kagan RM, Karalius B, Traite S, Meyer WA 3rd, Tassiopoulos KK, Seage GR 3rd, Seybolt LM, Burchett S, Hazra R; Pediatric HIV/AIDS Cohort Study (PHACS); Lurie RH, Yogev R, Sanders MA, Malee K, Hunter S, Shearer W, Paul M, Cooper N, Harris L, Purswani M, Baig M, Cintron A, Puga A, Navarro S, Garvie P, Blood J, Burchett S, Karthas N, Kammerer B, Wiznia A, Burey M, Nozyce M, Dieudonne A, Bettica L, Adubato S, Chen J, Bulkley MG, Ivey L, Grant M, Knapp K, Allison K, Wilkins M, Acevedo-Flores M, Rios H, Olivera V, Silio M, Jones M, Sirois P, Spector S, Norris K, Nichols S, McFarland E, Katai A, Dunn J, Paul S, Scott G, Bryan P, Willen E. Antiretroviral Drug Resistance Among Children and Youth in the United States With Perinatal HIV. Clin Infect Dis. 2016 Jul 1;63(1):133-137. doi: 10.1093/cid/ciw213. Epub 2016 Apr 7. PMID 27056398
- [Result] Van Dyke RB, Chadwick EG, Hazra R, Williams PL, Seage GR 3rd. The PHACS SMARTT Study: Assessment of the Safety of In Utero Exposure to Antiretroviral Drugs. Front Immunol. 2016 May 23;7:199. doi: 10.3389/fimmu.2016.00199. eCollection 2016. PMID 27242802
- [Result] Kacanek D, Malee K, Mellins CA, Tassiopoulos K, Smith R, Grant M, Lee S, Siddiqui DQ, Puga A. Exposure to Violence and Virologic and Immunological Outcomes Among Youth With Perinatal HIV in the Pediatric HIV/AIDS Cohort Study. J Adolesc Health. 2016 Jul;59(1):30-7. doi: 10.1016/j.jadohealth.2016.03.004. Epub 2016 Apr 15. PMID 27089837
- [Result] Moscicki AB, Yao TJ, Ryder MI, Russell JS, Dominy SS, Patel K, McKenna M, Van Dyke RB, Seage GR 3rd, Hazra R; Shiboski. The Burden of Oral Disease among Perinatally HIV-Infected and HIV-Exposed Uninfected Youth. PLoS One. 2016 Jun 14;11(6):e0156459. doi: 10.1371/journal.pone.0156459. eCollection 2016. PMID 27299992
- [Result] Spector SA, Brummel SS, Nievergelt CM, Maihofer AX, Singh KK, Purswani MU, Williams PL, Hazra R, Van Dyke R, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study (PHACS). Genetically determined ancestry is more informative than self-reported race in HIV-infected and -exposed children. Medicine (Baltimore). 2016 Sep;95(36):e4733. doi: 10.1097/MD.0000000000004733. PMID 27603370
- [Result] Lewis-de Los Angeles CP, Alpert KI, Williams PL, Malee K, Huo Y, Csernansky JG, Yogev R, Van Dyke RB, Sowell ER, Wang L; Pediatric HIV/AIDS Cohort Study (PHACS). Deformed Subcortical Structures Are Related to Past HIV Disease Severity in Youth With Perinatally Acquired HIV Infection. J Pediatric Infect Dis Soc. 2016 Dec;5(suppl 1):S6-S14. doi: 10.1093/jpids/piw051. PMID 27856671
- [Result] Sirois PA, Chernoff MC, Malee KM, Garvie PA, Harris LL, Williams PL, Woods SP, Nozyce ML, Kammerer BL, Yildirim C, Nichols SL; Memory and Executive Functioning Study of the Pediatric HIV/AIDS Cohort Study. Associations of Memory and Executive Functioning With Academic and Adaptive Functioning Among Youth With Perinatal HIV Exposure and/or Infection. J Pediatric Infect Dis Soc. 2016 Dec;5(suppl 1):S24-S32. doi: 10.1093/jpids/piw046. PMID 27856673
- [Result] Takemoto JK, Miller TL, Wang J, Jacobson DL, Geffner ME, Van Dyke RB, Gerschenson M; Pediatric HIVAIDS Cohort Study. Insulin resistance in HIV-infected youth is associated with decreased mitochondrial respiration. AIDS. 2017 Jan 2;31(1):15-23. doi: 10.1097/QAD.0000000000001299. PMID 27755108
- [Result] Uprety P, Patel K, Karalius B, Ziemniak C, Chen YH, Brummel SS, Siminski S, Van Dyke RB, Seage GR, Persaud D; Pediatric HIV/AIDS Cohort Study (PHACS). Human Immunodeficiency Virus Type 1 DNA Decay Dynamics With Early, Long-term Virologic Control of Perinatal Infection. Clin Infect Dis. 2017 Jun 1;64(11):1471-1478. doi: 10.1093/cid/cix192. PMID 28329153
- [Result] Lewis-de Los Angeles CP, Williams PL, Huo Y, Wang SD, Uban KA, Herting MM, Malee K, Yogev R, Csernansky JG, Nichols S, Van Dyke RB, Sowell ER, Wang L; Pediatric HIV/AIDS Cohort Study (PHACS) and the Pediatric Imaging, Neurocognition, and Genetics (PING) Study. Lower total and regional grey matter brain volumes in youth with perinatally-acquired HIV infection: Associations with HIV disease severity, substance use, and cognition. Brain Behav Immun. 2017 May;62:100-109. doi: 10.1016/j.bbi.2017.01.004. Epub 2017 Jan 10. PMID 28089557
- [Result] Neilan AM, Karalius B, Patel K, Van Dyke RB, Abzug MJ, Agwu AL, Williams PL, Purswani M, Kacanek D, Oleske JM, Burchett SK, Wiznia A, Chernoff M, Seage GR 3rd, Ciaranello AL; Pediatric HIV/AIDS Cohort Study and the International Maternal Adolescent and Pediatric AIDS Clinical Trials Network. Association of Risk of Viremia, Immunosuppression, Serious Clinical Events, and Mortality With Increasing Age in Perinatally Human Immunodeficiency Virus-Infected Youth. JAMA Pediatr. 2017 May 1;171(5):450-460. doi: 10.1001/jamapediatrics.2017.0141. PMID 28346597
- [Result] Shearer WT, Jacobson DL, Yu W, Siberry GK, Purswani M, Siminski S, Butler L, Leister E, Scott G, Van Dyke RB, Yogev R, Paul ME, Puga A, Colin AA, Kattan M; Pediatric HIV/AIDS Cohort Study. Long-term pulmonary complications in perinatally HIV-infected youth. J Allergy Clin Immunol. 2017 Oct;140(4):1101-1111.e7. doi: 10.1016/j.jaci.2017.01.031. Epub 2017 Mar 6. PMID 28279683
- [Result] Bellavia A, Williams PL, DiMeglio LA, Hazra R, Abzug MJ, Patel K, Jacobson DL, Van Dyke RB, Geffner ME; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) P219/219C Study, and the Pediatric HIV/AIDS Cohort Study (PHACS). Delay in sexual maturation in perinatally HIV-infected youths is mediated by poor growth. AIDS. 2017 Jun 1;31(9):1333-1341. doi: 10.1097/QAD.0000000000001486. PMID 28358737
- [Result] Jacobson DL, Stephensen CB, Miller TL, Patel K, Chen JS, Van Dyke RB, Mirza A, Schuster GU, Hazra R, Ellis A, Brummel SS, Geffner ME, Silio M, Spector SA, DiMeglio LA; Pediatric HIV/AIDS Cohort Study. Associations of Low Vitamin D and Elevated Parathyroid Hormone Concentrations With Bone Mineral Density in Perinatally HIV-Infected Children. J Acquir Immune Defic Syndr. 2017 Sep 1;76(1):33-42. doi: 10.1097/QAI.0000000000001467. PMID 28797019
- [Result] Garvie PA, Brummel SS, Allison SM, Malee KM, Mellins CA, Wilkins ML, Harris LL, Patton ED, Chernoff MC, Rutstein RM, Paul ME, Nichols SL; Pediatric HIV/AIDS Cohort Study. Roles of Medication Responsibility, Executive and Adaptive Functioning in Adherence for Children and Adolescents With Perinatally Acquired HIV. Pediatr Infect Dis J. 2017 Aug;36(8):751-757. doi: 10.1097/INF.0000000000001573. PMID 28709161
- [Result] Jao J, Yu W, Patel K, Miller TL, Karalius B, Geffner ME, DiMeglio LA, Mirza A, Chen JS, Silio M, McFarland EJ, Van Dyke RB, Jacobson D; Pediatric HIV/AIDS Cohort Study (PHACS) Adolescent Master Protocol (AMP) study. Improvement in lipids after switch to boosted atazanavir or darunavir in children/adolescents with perinatally acquired HIV on older protease inhibitors: results from the Pediatric HIV/AIDS Cohort Study. HIV Med. 2018 Mar;19(3):175-183. doi: 10.1111/hiv.12566. Epub 2017 Nov 21. PMID 29159965
- [Result] Harris LL, Chernoff MC, Nichols SL, Williams PL, Garvie PA, Yildirim C, McCauley SR, Woods SP; Memory and Executive Functioning Study of the Pediatric HIV/AIDS Cohort Study. Prospective memory in youth with perinatally-acquired HIV infection. Child Neuropsychol. 2018 Oct;24(7):938-958. doi: 10.1080/09297049.2017.1360854. Epub 2017 Aug 7. PMID 28782457
- [Result] Malee KM, Chernoff MC, Sirois PA, Williams PL, Garvie PA, Kammerer BL, Harris LL, Nozyce ML, Yildirim C, Nichols SL; Memory and Executive Functioning Study of the Pediatric HIV/AIDS Cohort Study. Impact of Perinatally Acquired HIV Disease Upon Longitudinal Changes in Memory and Executive Functioning. J Acquir Immune Defic Syndr. 2017 Aug 1;75(4):455-464. doi: 10.1097/QAI.0000000000001441. PMID 28481783
- [Result] Ryder MI, Yao TJ, Russell JS, Moscicki AB, Shiboski CH; Pediatric HIV/AIDS Cohort Study. Prevalence of periodontal diseases in a multicenter cohort of perinatally HIV-infected and HIV-exposed and uninfected youth. J Clin Periodontol. 2017 Jan;44(1):2-12. doi: 10.1111/jcpe.12646. Epub 2016 Nov 22. PMID 27801947
- [Result] Correia K, Williams PL. A hierarchical modeling approach for assessing the safety of exposure to complex antiretroviral drug regimens during pregnancy. Stat Methods Med Res. 2019 Feb;28(2):599-612. doi: 10.1177/0962280217732597. Epub 2017 Oct 3. PMID 28969502
- [Result] Williams PL, Jesson J. Growth and pubertal development in HIV-infected adolescents. Curr Opin HIV AIDS. 2018 May;13(3):179-186. doi: 10.1097/COH.0000000000000450. PMID 29432228
- [Result] Innes S, Patel K. Noncommunicable diseases in adolescents with perinatally acquired HIV-1 infection in high-income and low-income settings. Curr Opin HIV AIDS. 2018 May;13(3):187-195. doi: 10.1097/COH.0000000000000458. PMID 29432231
- [Result] Wilkinson JD, Williams PL, Yu W, Colan SD, Mendez A, Zachariah JPV, Van Dyke RB, Shearer WT, Margossian RE, Lipshultz SE; Pediatric HIV/AIDS Cohort Study (PHACS). Cardiac and inflammatory biomarkers in perinatally HIV-infected and HIV-exposed uninfected children. AIDS. 2018 Jun 19;32(10):1267-1277. doi: 10.1097/QAD.0000000000001810. PMID 29596110
- [Result] Starr JR, Huang Y, Lee KH, Murphy CM, Moscicki AB, Shiboski CH, Ryder MI, Yao TJ, Faller LL, Van Dyke RB, Paster BJ; Pediatric HIV/AIDS Cohort Study. Oral microbiota in youth with perinatally acquired HIV infection. Microbiome. 2018 May 31;6(1):100. doi: 10.1186/s40168-018-0484-6. PMID 29855347
- [Result] Alperen J, Davidson J, Siminski S, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study. Utility of the National Death Index in Identifying Deaths in a Clinic-Based, Multisite Cohort: The Experience of the Pediatric HIV/AIDS Cohort Study. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):e37-e39. doi: 10.1097/QAI.0000000000001763. No abstract available. PMID 29847477
- [Result] Collaborative Initiative for Paediatric HIV Education and Research (CIPHER) Global Cohort Collaboration; Slogrove AL, Schomaker M, Davies MA, Williams P, Balkan S, Ben-Farhat J, Calles N, Chokephaibulkit K, Duff C, Eboua TF, Kekitiinwa-Rukyalekere A, Maxwell N, Pinto J, Seage G 3rd, Teasdale CA, Wanless S, Warszawski J, Wools-Kaloustian K, Yotebieng M, Timmerman V, Collins IJ, Goodall R, Smith C, Patel K, Paul M, Gibb D, Vreeman R, Abrams EJ, Hazra R, Van Dyke R, Bekker LG, Mofenson L, Vicari M, Essajee S, Penazzato M, Anabwani G, Q Mohapi E, N Kazembe P, Hlatshwayo M, Lumumba M, Goetghebuer T, Thorne C, Galli L, van Rossum A, Giaquinto C, Marczynska M, Marques L, Prata F, Ene L, Okhonskaia L, Rojo P, Fortuny C, Naver L, Rudin C, Le Coeur S, Volokha A, Rouzier V, Succi R, Sohn A, Kariminia A, Edmonds A, Lelo P, Ayaya S, Ongwen P, Jefferys LF, Phiri S, Mubiana-Mbewe M, Sawry S, Renner L, Sylla M, Abzug MJ, Levin M, Oleske J, Chernoff M, Traite S, Purswani M, Chadwick EG, Judd A, Leroy V. The epidemiology of adolescents living with perinatally acquired HIV: A cross-region global cohort analysis. PLoS Med. 2018 Mar 1;15(3):e1002514. doi: 10.1371/journal.pmed.1002514. eCollection 2018 Mar. PMID 29494593
- [Result] Margossian R, Williams PL, Yu W, Jacobson DL, Geffner ME, DiMeglio LA, Van Dyke RB, Spector SA, Schuster GU, Stephensen CB, Miller TL, Lipshultz SE; Pediatric HIV/AIDS Cohort Study (PHACS). Markers of Bone Mineral Metabolism and Cardiac Structure and Function in Perinatally HIV-Infected and HIV-Exposed but Uninfected Children and Adolescents. J Acquir Immune Defic Syndr. 2019 Jun 1;81(2):238-246. doi: 10.1097/QAI.0000000000002007. PMID 30865170
- [Result] Smith R, Huo Y, Tassiopoulos K, Rutstein R, Kapetanovic S, Mellins C, Kacanek D, Malee K; Pediatric HIV/AIDS Cohort Study (PHACS). Mental Health Diagnoses, Symptoms, and Service Utilization in US Youth with Perinatal HIV Infection or HIV Exposure. AIDS Patient Care STDS. 2019 Jan;33(1):1-13. doi: 10.1089/apc.2018.0096. PMID 30601062
- [Result] Lee KH, Coull BA, Moscicki AB, Paster BJ, Starr JR. Bayesian variable selection for multivariate zero-inflated models: Application to microbiome count data. Biostatistics. 2020 Jul 1;21(3):499-517. doi: 10.1093/biostatistics/kxy067. PMID 30590511
- [Result] Shiboski CH, Yao TJ, Russell JS, Ryder MI, Van Dyke RB, Seage GR 3rd, Moscicki AB; Pediatric HIV/AIDS Cohort Study. The association between oral disease and type of antiretroviral therapy among perinatally HIV-infected youth. AIDS. 2018 Nov 13;32(17):2497-2505. doi: 10.1097/QAD.0000000000001965. PMID 30096069
- [Result] Williams PL, Correia K, Karalius B, Van Dyke RB, Wilkinson JD, Shearer WT, Colan SD, Lipshultz SE; Pediatric HIV/AIDS Cohort Study. Cardiac status of perinatally HIV-infected children: assessing combination antiretroviral regimens in observational studies. AIDS. 2018 Oct 23;32(16):2337-2346. doi: 10.1097/QAD.0000000000001988. PMID 30102660
- [Result] Moscicki AB, Karalius B, Tassiopoulos K, Yao TJ, Jacobson DL, Patel K, Purswani M, Seage GR; Pediatric HIV/AIDS Cohort Study. Human Papillomavirus Antibody Levels and Quadrivalent Vaccine Clinical Effectiveness in Perinatally Human Immunodeficiency Virus-infected and Exposed, Uninfected Youth. Clin Infect Dis. 2019 Sep 13;69(7):1183-1191. doi: 10.1093/cid/ciy1040. PMID 30927547
- [Result] Yildirim C, Garvie PA, Chernoff M, Wilkins ML, Patton ED, Williams PL, Nichols SL; Memory and Executive Functioning Study of the Pediatric HIV/AIDS Cohort Study. The Role of Pharmacy Refill Measures in Assessing Adherence and Predicting HIV Disease Markers in Youth with Perinatally-Acquired HIV (PHIV). AIDS Behav. 2019 Aug;23(8):2109-2120. doi: 10.1007/s10461-019-02468-x. PMID 30929147
- [Result] Collaborative Initiative for Paediatric HIV Education and Research (CIPHER) Global Cohort Collaboration. Incidence of switching to second-line antiretroviral therapy and associated factors in children with HIV: an international cohort collaboration. Lancet HIV. 2019 Feb;6(2):e105-e115. doi: 10.1016/S2352-3018(18)30319-9. PMID 30723008
- [Result] Moscicki AB, Yao TJ, Russell JS, Farhat S, Scott M, Magpantay L, Halec G, Shiboski CH, Ryder MI; Pediatric HIV/AIDS Cohort Study. Biomarkers of oral inflammation in perinatally HIV-infected and perinatally HIV-exposed, uninfected youth. J Clin Periodontol. 2019 Nov;46(11):1072-1082. doi: 10.1111/jcpe.13179. Epub 2019 Sep 5. PMID 31385616
- [Result] Ryder MI, Shiboski C, Yao TJ, Moscicki AB. Current trends and new developments in HIV research and periodontal diseases. Periodontol 2000. 2020 Feb;82(1):65-77. doi: 10.1111/prd.12321. PMID 31850628
- [Result] Bather JR, Williams PL, Broadwell C, Smith R, Patel K, Garvie PA, Karalius B, Kacanek D, Mellins CA, Malee K; Pediatric HIV/AIDS Cohort Study (PHACS). Racial/Ethnic Disparities in Longitudinal Emotional-Behavioral Functioning Among Youth Born to Women Living With HIV. J Acquir Immune Defic Syndr. 2021 Jul 1;87(3):889-898. doi: 10.1097/QAI.0000000000002665. PMID 33675617
- [Result] Dirajlal-Fargo S, Williams PL, Broadwell C, McFarland EJ, Powis KM, Jacobson DL, Jao J; Pediatric HIV/AIDS Cohort Study (PHACS). Brief Report: Youth Living With Perinatally Acquired HIV Have Lower Physical Activity Levels as They Age Compared With HIV-Exposed Uninfected Youth. J Acquir Immune Defic Syndr. 2021 May 1;87(1):700-705. doi: 10.1097/QAI.0000000000002622. PMID 33443964
- [Result] Nichols SL, Brummel S, Malee KM, Mellins CA, Moscicki AB, Smith R, Cuadra AM, Bryant K, Boyce CA, Tassiopoulos KK; Pediatric HIV/AIDS Cohort Study. The Role of Behavioral and Neurocognitive Functioning in Substance Use Among Youth with Perinatally Acquired HIV Infection and Perinatal HIV Exposure Without Infection. AIDS Behav. 2021 Sep;25(9):2827-2840. doi: 10.1007/s10461-021-03174-3. Epub 2021 Feb 22. PMID 33616833
- [Result] Shiau S, Brummel SS, Kennedy EM, Hermetz K, Spector SA, Williams PL, Kacanek D, Smith R, Drury SS, Agwu A, Ellis A, Patel K, Seage GR 3rd, Van Dyke RB, Marsit CJ; Pediatric HIV/AIDS Cohort Study (PHACS). Longitudinal changes in epigenetic age in youth with perinatally acquired HIV and youth who are perinatally HIV-exposed uninfected. AIDS. 2021 Apr 1;35(5):811-819. doi: 10.1097/QAD.0000000000002805. PMID 33587437
- [Result] Schulte F, King OD, Paster BJ, Moscicki AB, Yao TJ, Van Dyke RB, Shiboski C, Ryder M, Seage G, Hardt M; Pediatric HIV/AIDS Cohort Study. Salivary metabolite levels in perinatally HIV-infected youth with periodontal disease. Metabolomics. 2020 Sep 11;16(9):98. doi: 10.1007/s11306-020-01719-6. PMID 32915320
- [Result] Jacobson DL, Yu W, Hazra R, Brummel S, Geffner ME, Patel K, Borkowsky W, Wang J, Chen JS, Mirza A, DiMeglio LA; Pediatric HIV/AIDS Cohort Study. Fractures in children and adolescents living with perinatally acquired HIV. Bone. 2020 Oct;139:115515. doi: 10.1016/j.bone.2020.115515. Epub 2020 Jun 30. PMID 32619695
- [Result] Gojanovich GS, Jacobson DL, Jao J, Russell JS, Van Dyke RB, Libutti DE, Sharma TS, Geffner ME, Gerschenson M. Mitochondrial Dysfunction and Insulin Resistance in Pubertal Youth Living with Perinatally Acquired HIV. AIDS Res Hum Retroviruses. 2020 Sep;36(9):703-711. doi: 10.1089/AID.2020.0067. Epub 2020 Jul 20. PMID 32586116
- [Result] Lewis-de Los Angeles CP, Williams PL, Jenkins LM, Huo Y, Malee K, Alpert KI, Uban KA, Herting MM, Csernansky JG, Nichols SL, Van Dyke RB, Sowell ER, Wang L; Pediatric HIV/AIDS Cohort Study (PHACS) and the Pediatric Imaging, Neurocognition, and Genetics (PING) Study. Brain morphometric differences in youth with and without perinatally-acquired HIV: A cross-sectional study. Neuroimage Clin. 2020;26:102246. doi: 10.1016/j.nicl.2020.102246. Epub 2020 Mar 16. PMID 32251906
- [Result] McManus M, Karalius B, Patel K, Persaud D, Luzuriaga K; Pediatric HIV/AIDS Cohort Study. Quantitative HIV-1-specific antibodies as predictors of peripheral blood cell-associated HIV-1 DNA concentrations. AIDS. 2020 Jul 1;34(8):1117-1126. doi: 10.1097/QAD.0000000000002525. PMID 32287055
- [Result] Attia EF, Jacobson D, Yu W, Crowell CS, Maleche-Obimbo E, Williams PL, West TE, Burchett SK, Kattan M, Colin AA, Eskander S, Chung MH, Crothers K, Shearer WT; Pediatric HIV/AIDS Cohort Study. Immune imbalance and activation are associated with lower lung function in youth with perinatally acquired HIV. J Allergy Clin Immunol. 2020 May;145(5):1473-1476. doi: 10.1016/j.jaci.2019.12.890. Epub 2019 Dec 23. PMID 31874184
- [Result] Garvie PA, Nichols SL, Williams PL, Harris LL, Kammerer B, Chernoff MC, Figueroa V, Woods SP. Development and reliability of the Prospective Memory Assessment for Children & Youth (PROMACY): A preliminary study in a nonclinical sample. Appl Neuropsychol Child. 2019 Oct-Dec;8(4):333-346. doi: 10.1080/21622965.2018.1486194. Epub 2018 Oct 8. PMID 30295555
- [Result] Geffner ME, Patel K, Jacobson DL, Wu J, Miller TL, Hazra R, Gerschenson M, Sharma T, Silio M, Jao J, Takemoto JK, Van Dyke RB, DiMeglio LA; Pediatric HIV/AIDS Cohort Study (PHACS). Changes in insulin sensitivity over time and associated factors in HIV-infected adolescents. AIDS. 2018 Mar 13;32(5):613-622. doi: 10.1097/QAD.0000000000001731. PMID 29280758
- [Result] Fulcher IR, Tchetgen Tchetgen EJ, Williams PL. Mediation Analysis for Censored Survival Data Under an Accelerated Failure Time Model. Epidemiology. 2017 Sep;28(5):660-666. doi: 10.1097/EDE.0000000000000687. PMID 28574921
- [Result] Hermetet-Lindsay KD, Correia KF, Williams PL, Smith R, Malee KM, Mellins CA, Rutstein RM; Pediatric HIV/AIDS Cohort Study. Contributions of Disease Severity, Psychosocial Factors, and Cognition to Behavioral Functioning in US Youth Perinatally Exposed to HIV. AIDS Behav. 2017 Sep;21(9):2703-2715. doi: 10.1007/s10461-016-1508-5. PMID 27475941
- [Result] Redmond SM, Yao TJ, Russell JS, Rice ML, Hoffman HJ, Siberry GK, Frederick T, Purswani M, Williams PL; Pediatric HIV/AIDS Cohort Study. Longitudinal Evaluation of Language Impairment in Youth With Perinatally Acquired Human Immunodeficiency Virus (HIV) and Youth With Perinatal HIV Exposure. J Pediatric Infect Dis Soc. 2016 Dec;5(suppl 1):S33-S40. doi: 10.1093/jpids/piw045. PMID 27856674
- [Result] Nichols SL, Chernoff MC, Malee KM, Sirois PA, Woods SP, Williams PL, Yildirim C, Delis D, Kammerer B; Memory and Executive Functioning Study of the Pediatric HIV/AIDS Cohort Study. Executive Functioning in Children and Adolescents With Perinatal HIV Infection and Perinatal HIV Exposure. J Pediatric Infect Dis Soc. 2016 Dec;5(suppl 1):S15-S23. doi: 10.1093/jpids/piw049. PMID 27856672
- [Result] Malee KM, Smith RA, Mellins CA; Pediatric HIV/AIDS Cohort Study. Brain and Cognitive Development Among U.S. Youth With Perinatally Acquired Human Immunodeficiency Virus Infection. J Pediatric Infect Dis Soc. 2016 Dec;5(suppl 1):S1-S5. doi: 10.1093/jpids/piw041. No abstract available. PMID 27856670
- [Result] Purswani MU, Karalius B, Yao TJ, Schmid DS, Burchett SK, Siberry GK, Patel K, Van Dyke RB, Yogev R; Pediatric HIV/AIDS Cohort Study (PHACS); Lurie RH, Yogev R, Sanders MA, Malee K, Hunter S, Shearer W, Paul M, Cooper N, Harris L, Purswani M, Baig M, Cintron A, Puga A, Navarro S, Garvie P, Blood J, Burchett S, Karthas N, Kammerer B, Wiznia A, Burey M, Nozyce M, Dieudonne A, Bettica L, Adubato S, Chen J, Bulkley MG, Ivey L, Grant M, Knapp K, Allison K, Wilkins M, Acevedo-Flores M, Rios H, Olivera V, Silio M, Jones M, Sirois P, Spector S, Norris K, Nichols S, McFarland E, Katai A, Dunn J, Paul S, Scott G, Bryan P, Willen E. Prevalence and Persistence of Varicella Antibodies in Previously Immunized Children and Youth With Perinatal HIV-1 Infection. Clin Infect Dis. 2016 Jan 1;62(1):106-114. doi: 10.1093/cid/civ734. Epub 2015 Sep 18. PMID 26385992
- [Result] Koller M, Patel K, Chi BH, Wools-Kaloustian K, Dicko F, Chokephaibulkit K, Chimbetete C, Avila D, Hazra R, Ayaya S, Leroy V, Truong HK, Egger M, Davies MA; IeDEA, NISDI, PHACS and IMPAACT 219C studies. Immunodeficiency in children starting antiretroviral therapy in low-, middle-, and high-income countries. J Acquir Immune Defic Syndr. 2015 Jan 1;68(1):62-72. doi: 10.1097/QAI.0000000000000380. PMID 25501345
- [Result] Berman CA, Kacanek D, Nichamin M, Wilson D, Davtyan M, Salomon L, Patel K, Reznick M, Tassiopoulos K, Lee S, Bauermeister J, Paul M, Aldape T, Seage Iii GR. Using Social Media and Technology to Communicate in Pediatric HIV Research: Qualitative Study With Young Adults Living With or Exposed to Perinatal HIV. JMIR Pediatr Parent. 2020 Jun 23;3(1):e20712. doi: 10.2196/20712. PMID 32540839
- [Result] Moscicki AB, Farhat S, Yao TJ, Ryder MI, Russell JS, Van Dyke RB, Hazra R, Shiboski CH; Pediatric HIVAIDS Cohort Study. Oral Human Papillomavirus in Youth From the Pediatric HIV/AIDS Cohort Study. Sex Transm Dis. 2016 Aug;43(8):498-500. doi: 10.1097/OLQ.0000000000000495. PMID 27414680
- [Result] Jao J, Jacobson DL, Russell JS, Wang J, Yu W, Gojanovich GS, Siminski S, Hyzy L, Geffner ME, Gerschenson M; for the Pediatric HIV/AIDS Cohort Study. Perinatally acquired HIV infection is associated with abnormal blood mitochondrial function during childhood/adolescence. AIDS. 2021 Jul 15;35(9):1385-1394. doi: 10.1097/QAD.0000000000002884. PMID 33730749
- [Result] Rawat P, Brummel SS, Singh KK, Kim J, Frazer KA, Nichols S, Seage GR, Williams PL, Van Dyke RB, Harismendy O, Trout RN, Spector SA. Genomics Links Inflammation With Neurocognitive Impairment in Children Living With Human Immunodeficiency Virus Type-1. J Infect Dis. 2021 Sep 1;224(5):870-880. doi: 10.1093/infdis/jiaa792. PMID 33373444
- [Result] Barnard-Mayers R, Kouser H, Cohen JA, Tassiopoulos K, Caniglia EC, Moscicki AB, Campos NG, Caunca MR, Seage GRS, Murray EJ. A case study and proposal for publishing directed acyclic graphs: The effectiveness of the quadrivalent human papillomavirus vaccine in perinatally HIV Infected girls. J Clin Epidemiol. 2022 Apr;144:127-135. doi: 10.1016/j.jclinepi.2021.12.028. Epub 2022 Jan 5. PMID 34998951
- [Result] Collaborative Initiative for Paediatric HIV Education and Research (CIPHER) Global Cohort Collaboration; Jesson J, Crichton S, Quartagno M, Yotebieng M, Abrams EJ, Chokephaibulkit K, Le Coeur S, Ake-Assi MH, Patel K, Pinto J, Paul M, Vreeman R, Davies MA, Ben-Farhat J, Van Dyke R, Judd A, Mofenson L, Vicari M, Seage G 3rd, Bekker LG, Essajee S, Gibb D, Penazzato M, Collins IJ, Wools-Kaloustian K, Slogrove A, Powis K, Williams P, Matshaba M, Thahane L, Nyasulu P, Lukhele B, Mwita L, Kekitiinwa-Rukyalekere A, Wanless S, Goetghebuer T, Thorne C, Warszawski J, Galli L, van Rossum AMC, Giaquinto C, Marczynska M, Marques L, Prata F, Ene L, Okhonskaya L, Navarro M, Frick A, Naver L, Kahlert C, Volokha A, Chappell E, Pape JW, Rouzier V, Marcelin A, Succi R, Sohn AH, Kariminia A, Edmonds A, Lelo P, Lyamuya R, Ogalo EA, Odhiambo FA, Haas AD, Bolton C, Muhairwe J, Tweya H, Sylla M, D'Almeida M, Renner L, Abzug MJ, Oleske J, Purswani M, Teasdale C, Nuwagaba-Biribonwoha H, Goodall R, Leroy V. Growth and CD4 patterns of adolescents living with perinatally acquired HIV worldwide, a CIPHER cohort collaboration analysis. J Int AIDS Soc. 2022 Mar;25(3):e25871. doi: 10.1002/jia2.25871. PMID 35255197
- [Result] Dirajlal-Fargo S, Jacobson DL, Yu W, Mirza A, Geffner ME, Jao J, McComsey GA. Gut Dysfunction Markers Are Associated With Body Composition in Youth Living With Perinatally Acquired Human Immunodeficiency Virus. Clin Infect Dis. 2022 Sep 29;75(6):945-952. doi: 10.1093/cid/ciac053. PMID 35090002
- [Result] Shiau S, Yu W, Jacobson DL, Nichols S, McFarland EJ, Chen JS, Dirajlal-Fargo S, Surowiec K, Geffner ME, Jao J; Pediatric HIV/AIDS Cohort Study. Components of metabolic syndrome associated with lower neurocognitive performance in youth with perinatally acquired HIV and youth who are HIV-exposed uninfected. J Neurovirol. 2021 Oct;27(5):702-715. doi: 10.1007/s13365-021-01005-8. Epub 2021 Sep 15. PMID 34524627
- [Result] Brummel SS, Van Dyke RB, Patel K, Purswani M, Seage GR, Yao TJ, Hazra R, Karalius B, Williams PL; Pediatric HIV/AIDS Cohort Study. Analyzing Longitudinally Collected Viral Load Measurements in Youth With Perinatally Acquired HIV Infection: Problems and Possible Remedies. Am J Epidemiol. 2022 Sep 28;191(10):1820-1830. doi: 10.1093/aje/kwac125. PMID 35872591
- [Result] Sirois PA, Huo Y, Nozyce ML, Garvie PA, Harris LL, Malee K, McEvoy R, Mellins CA, Nichols SL, Smith R, Tassiopoulos K; Pediatric HIV/AIDS Cohort Study. Ageing with HIV: a longitudinal study of markers of resilience in young adults with perinatal exposure to HIV, with or without perinatally acquired HIV. J Int AIDS Soc. 2022 Sep;25 Suppl 4(Suppl 4):e25982. doi: 10.1002/jia2.25982. PMID 36176020
- [Result] Lemon TL, Tassiopoulos K, Tsai AC, Cantos K, Escudero D, Quinn MK, Kacanek D, Berman C, Salomon L, Nichols S, Chadwick EG, Seage GR 3rd, Williams PL; Pediatric HIV/AIDS Cohort Study (PHACS). Health Insurance Coverage, Clinical Outcomes, and Health-Related Quality of Life Among Youth Born to Women Living With HIV. J Acquir Immune Defic Syndr. 2023 Jan 1;92(1):6-16. doi: 10.1097/QAI.0000000000003100. PMID 36150048
- [Result] Global variations in pubertal growth spurts in adolescents living with perinatal HIV. AIDS. 2023 Aug 1;37(10):1603-1615. doi: 10.1097/QAD.0000000000003602. Epub 2023 May 17. PMID 37204259
- [Result] Caceres GA, Scambray KA, Malee K, Smith R, Williams PL, Wang L, Jenkins LM; Pediatric HIV/AIDS Cohort Study. Relationship between brain structural network integrity and emotional symptoms in youth with perinatally-acquired HIV. Brain Behav Immun. 2024 Feb;116:101-113. doi: 10.1016/j.bbi.2023.11.026. Epub 2023 Dec 2. PMID 38043871
- [Result] Dirajlal-Fargo S, Jacobson DL, Yu W, Mirza A, Geffner ME, Mccomsey GA, Jao J; Pediatric HIV/AIDS Cohort Study (PHACS). Longitudinal changes in body fat and metabolic complications in young people with perinatally acquired HIV. HIV Med. 2024 Feb;25(2):233-244. doi: 10.1111/hiv.13566. Epub 2023 Oct 16. PMID 37845017
- [Result] Dirajlal-Fargo S, Yu W, Jacobson DL, Mirza A, Geffner ME, Jao J, McComsey GA; Pediatric HIV/AIDS Cohort Study (PHACS). Gut permeability is associated with lower insulin sensitivity in youth with perinatally acquired HIV. AIDS. 2024 Jul 1;38(8):1163-1171. doi: 10.1097/QAD.0000000000003896. Epub 2024 Mar 28. PMID 38564437
- [Result] Gojanovich GS, Yu W, Zhang ZJ, Jacobson DL, Yao TJ, Jao J, Libutti DE, Geffner ME, Gerschenson M; Pediatric HIV/AIDS Cohort Study. Longitudinal changes in mitochondrial-associated measures and insulin resistance in youth with perinatally-acquired HIV in the U.S. Mitochondrion. 2024 Sep;78:101936. doi: 10.1016/j.mito.2024.101936. Epub 2024 Jul 14. PMID 39009104
- [Result] DiMeglio LA, Yu W, Kalkwarf HJ, Brummel S, Chen JS, Geffner ME, McFarland EJ, Mirza A, Patel K, Shiau S, Jacobson DL; Pediatric HIV/AIDS Cohort Study. Bone Accrual Trajectories in Children and Adolescents With Perinatal HIV Infection. J Clin Endocrinol Metab. 2025 May 19;110(6):e1783-e1792. doi: 10.1210/clinem/dgae631. PMID 39312415
- See also: Pediatric HIV/AIDS Cohort Study — https://phacsstudy.org